CLINICAL TRIAL: NCT03588130
Title: A Multicenter , Prospective, Randomized, Placebo Controlled, Adaptive Design Study Performed to Evaluate the Safety and the Efficacy of EscharEx (EX-02 Formulation) in Debridement of Venous Leg Ulcers
Brief Title: A Study to Evaluate the Safety and the Efficacy of EscharEx (EX-02 Formulation) in Debridement of Venous Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW2017-06-28
Record Dates: First submitted 2018-06-20; First posted 2018-07-17 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-01

CONDITIONS: Venous Leg Ulcer
Keywords: Debridement
MeSH Terms: conditions — Varicose Ulcer | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of subjects, study team on sites (e.g. investigators, study nurses etc.) and sponsor team to the assigned treatment will be employed between EX-02 arm and Gel Vehicle arm. Since the NSSOC appearance and dosing regimen are different from that of IMP (EX-02 or Gel vehicle), treatment with NSSOC arm can not be masked to study team or sponsor.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EscharEx (5% EX-02 formulation) (Active Comparator): Debridement will be performed with 5% EX-02 for 24±3 hours, up to 8 applications
  Interventions: Drug: EscharEx (5% EX-02 formulation)
- Gel Vehicle (Placebo Comparator): Debridement will be performed with Gel vehicle for 24±3 hours, up to 8 applications
  Interventions: Drug: Gel Vehicle
- Non-surgical standard of care (NSSOC) (Active Comparator): Debridement will be performed with NSSOC (Santyl or commercially approved Hydrogel) per routine procedures, until complete debridement is achieved
  Interventions: Drug: Non-surgical standard of care (NSSOC)

INTERVENTIONS:
Drug: EscharEx (5% EX-02 formulation) — Active arm
  Arms: EscharEx (5% EX-02 formulation)
Drug: Gel Vehicle — Control arm
  Arms: Gel Vehicle
Drug: Non-surgical standard of care (NSSOC) — Santyl (Enzymatic debridement) or commercially approved Hydrogel
  Arms: Non-surgical standard of care (NSSOC)

SUMMARY:
This study is a multicenter, prospective, randomized, placebo controlled, adaptive design study performed to assess the safety and the efficacy of 5% EscharEx (EX-02) compared to Gel Vehicle (placebo) and non-surgical standard of care (NSSOC), in debridement of Venous Leg Ulcers (VLU) (in a ratio of 2:2:1) in debridement of VLU.

The main objective of this study is:

To assess the safety and the efficacy of EscharEx (EX-02 formulation) compared to Gel Vehicle (placebo) and non-surgical standard of care (NSSOC), in debridement of Venous Leg Ulcers (VLU).

120 randomized adult patients with VLU that fail to heal for 4 weeks to 2 years, and with >50% non-viable tissue (necrotic/slough/fibrin) on the VLU. The maximum number of patients to be enrolled is 160.

The total duration of the study of each participating subject is up to 17 weeks: screening (1 week) + Daily visit period (up to 2 weeks) + Twice-weekly visits period (2 weeks) + Weekly visits period (10 weeks) + closure confirmation (up to 2 weeks, if applicable).

Each patient will go through 4 periods during the trial:

1. Screening period (2 visits, 7 [+2] days apart). Including: recording demographics, medical history and concomitant medications, vital signs, physical examination, clinical laboratory tests, wound photography and assessments and questionnaires (pain, wound status and QoL). During this period, wounds will be treated by standard treatment (e.g. appropriate dressing, compression bandage) per investigator discretion, with the exclusion of mechanical and surgical debridement.

   During the one week screening period, patients whose wound size (surface area, as measured by eKare inSightTM) decreases by more than 20 percent will be excluded.
2. Daily visits period (up to 8 daily site visits within up to 14 days): During the Daily visit period, the patient will arrive daily to site visits. During each visit, adverse events, concomitant medication, vital signs and pain will be recorded, the wound will be washed, photographed and assessed for wound size (by eKare inSightTM), % of non viable tissue (by clinical assessment), and wound healing status (assessed clinically).

   Eligible patients will be randomized into one of the study arms: EX-02, or Gel Vehicle (Placebo), or NSSOC in a 2:2:1 ratio. Patients will be treated with up to 8 daily 24±3 hours applications or until complete debridement is achieved, whichever occurs first.

   On the weekends between treatments of EX-02 or Gel material, the wound will be dressed with a compatible dressing, and by compression therapy. Patients treated with NSSOC continue using NSSOC during the weekend according to label or instructions for use, and compression therapy.
3. Twice-weekly visits period (4 visits within 14 days): the patients will be followed twice weekly for two weeks, (4 visits within 14 days). During each visit, safety parameters will be recorded (AEs, concomitant medications, pain, vital signs), the wound will be washed, photographed and assessed for wound size (by eKare inSightTM), % of nonviable tissue (by clinical assessment), and wound healing status (assessed clinically).

   The investigator will clinically assess complete debridement, upon achieving a viable wound bed after removal of all non-viable tissue, suitable for initiation of the wound healing stage.
4. Weekly visits period (up to10 visits within up to 10 weeks): patients will be followed once weekly for 10 weeks or until complete wound closure was achieved, (up to10 visits within up to 10 weeks). During each weekly visit, safety parameters will be recorded (AEs, concomitant medications, pain, vital signs), the wound will be washed, photographed and assessed for wound size (by eKare inSightTM), % of nonviable tissue (by clinical assessment), and wound healing status (assessed clinically).

The investigator will clinically assess complete debridement, upon achieving a viable wound bed after removal of all non-viable tissue, suitable for initiation of the wound healing stage.

Complete wound closure defined as skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits, 2 weeks apart will be assessed clinically. Thus, if closure occurs close to the end of weekly visit period, i.e. on 9th or 10th visit of the weekly period, an additional confirmation visit will be performed 2 weeks later.

ELIGIBILITY:
Inclusion Criteria

1. Patients, men or women, between 18 and 90 years of age,
2. Patients with a VLU (determined by medical history, physical examination, and an ultrasound scan demonstrating venous insufficiency),
3. Wound is present for at least 4 weeks but no longer than 2 years.
4. The necrotic/slough/fibrin non-viable tissue area is at least 50% of wound area (assessed by clinical evaluation),
5. Target wound surface area is in the range of 2-100 cm2 (assessed by eKare inSightTM),
6. Patient understands the nature of the procedure, is able to adhere to the protocol regimen, and provides a written informed consent prior to any study procedure.

Exclusion Criteria

1. Wound size decreased by > 20% after 1 week of standard-of-care-only period (screening period),
2. Patients with more than one leg ulcer, on the leg of the target wound, with an area greater than or equal to 2cm2,
3. Signs of clinically significant infection including purulent discharge, deep-tissue abscess, erysipelas, cellulitis, etc.,
4. Severely damaged skin (e.g. abrasion, exfoliation) extending >2 cm around the wound's edge,
5. Presence of gangrene, signs of systemic infection, sepsis, or osteomyelitis during screening phase,
6. Clinical suspicion of skin cancer (e.g. BCC, SCC, melanoma, sarcoma), which was not ruled out by biopsy,
7. Patients with skin disorders unrelated to the wound that are presented adjacent to the wound,
8. Patients suffering from chronic skin disorders (Idiopathic Pruritus, Psoriasis, Panniculitis, Pyoderma Gangrenosum, etc.) that might deteriorate as a result of local trauma or debridement,
9. Wound has sinus tracts or tunnels extending under healthy tissue (following debridement "un-roofing"- if relevant), or penetrating into joint capsule,
10. Vascular operations in proximity to the wound in the last month,
11. Patients with primary lymphatic edema,
12. A significant decrease in the arterial blood flow of the extremity
13. Patients with pre-enrolment wounds which are covered by eschar heavily saturated with iodine or by silver sulfadiazine (SSD) pseudoeschar (i.e. pseudoeschar as a result of SSD treatment),
14. History of allergy or atopic disease or a known sensitivity to pineapples, papaya, bromelain or papain, as well as known sensitivity to latex proteins (known as latex-fruit syndrome), bee venom or olive tree pollen,
15. Patients with poor nutritional status: albumin < 2.5g/dl, poorly controlled Diabetes Mellitus (for diabetic patients; HbA1c > 12%), anemia (hemoglobin<8 g/dL), a leukocyte counts < 3,800// μl or >15000/μl, platelets <100,000/μl, abnormal liver function (AST, ALT>2 x upper limit of normal range), renal failure (Cr > 2.5 mg/dl), BMI>48,
16. Patients undergoing renal or peritoneal dialysis,
17. Any condition that would preclude safe participation in the study, e.g. evidence of significant or unstable cardiovascular, pulmonary, liver, hematological, immunological, or neoplastic disease, or any immediate life threatening condition,
18. Recent history (less than 6 months) of myocardial infarction (MI) or concurrent acute injury or disease that might compromise the patient's welfare,
19. Patient is currently receiving, or has received at any time within three months prior to enrollment, any medications or treatments known to affect the wound healing processes; these include, chronic systemic steroid intake with topical skin changes (i.e. thin, fragile skin with multiple heamatomas or previous laceration history) immuno-suppressive drugs, radiation therapy, immunomodulating medications and chemotherapy,
20. Mentally incapacitated adults who are incapable of giving legal consent (e.g. dementia, psychiatric patients, etc.),
21. Concurrent use of non-approved drugs or alcohol abuse,
22. Pregnant women (positive pregnancy test) or nursing mothers,
23. Exposure to investigational intervention within three months prior to enrollment, or anticipated participation in another investigational drug trial or other intervention trial, while enrolled in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of complete debridement in EX-02 vs. Gel Vehicle arms, scored dichotomously (yes/no), clinically assessed | up to 8 applications, within 14 days
  The clinical assessor will define complete debridement, after each application during the daily visits period

CONTACTS AND LOCATIONS:
Locations (22):
- United States (21):
  - ILD Research Center, Carlsbad, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Felix Sigal. D.P.M, PC, Los Angeles, California
  - Stanford, Redwood City, California
  - Center for Clinical Research Inc., San Francisco, California
  - Medstar Health Georgetown University, Washington D.C., District of Columbia
  - C & R Research Services USA, Inc, Coral Gables, Florida
  - INTEGRAL - Clinical Trials Solutions, Doral, Florida
  - University of Miami, Miami, Florida
  - Barry University Clinical Research, Miami Beach, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center/Boston University Medical Center, Boston, Massachusetts
  - South Shore Health System, Center for Wound Healing, Weymouth, Massachusetts
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Atlantic Health System - Overlook Wound Care Center, Summit, New Jersey
  - Bey Lea Ambulatory Surgical Center, Toms River, New Jersey
  - NYU Winthrop Hospital, Mineola, New York
  - Mount Sinai St. Luke's Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - AZH Wound Center, Milwaukee, Wisconsin
- Hopitaux Universitaires de Geneva, Geneva, Canton, Switzerland

REFERENCES:
- [Derived] Shoham Y, Snyder RJ, Katz Levy Y, David Zarbiv K, Klinger E, Kramer M, Dove CR, Avrahami R, Reyzelman A, Sigal F, Tovmassian G, Shapira E, Harats M, Perez-Clavijo F, Lantis JC, Cazzell SM, Dhillon YS, Cuffy CA, Egozi D, Vayser D, Singer AJ, Galperin RC, Hanft JR, Martinez C, Shalom A, Toutous-Trellu L, Rosenberg L. Once daily Bromelain-based enzymatic debridement of venous leg ulcers versus gel vehicle (placebo) and non-surgical standard of care: a three-arm multicenter, double blinded, randomized controlled study. EClinicalMedicine. 2024 Jul 27;75:102750. doi: 10.1016/j.eclinm.2024.102750. eCollection 2024 Sep. PMID 39763591